CLINICAL TRIAL: NCT00937573
Title: Xience V at WFUBMC: Real World Outcomes Using Second Generation DES
Brief Title: Xience V at Wake Forest University Baptist Medical Center (WFUBMC)
Status: Completed | Type: Observational
Sponsor: Wake Forest University (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Other Study IDs: ACS-6814
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2014-12

CONDITIONS: Percutaneous Coronary Intervention; Stents
Keywords: stents; mortality; revascularization; stent thrombosis; Drug-Eluting Stents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Xience V: Percutaneous coronary intervention with Xience V stent placement
- Historical BMS: Percutaneous coronary intervention with bare metal stent placement prior to availability of Cypher, Taxus, or Xience V drug eluting stents at WFUBMC
- Historical DES: Percutaneous coronary intervention with drug eluting stent placement prior to availability of Xience V drug eluting stents at WFUBMC
- Contemporary BMS: Percutaneous coronary intervention with bare metal stent placement after Xience V drug eluting stents were available for use at WFUBMC
- Contemporary DES: Percutaneous coronary intervention with Cypher or Taxus drug eluting stent placement after Xience V drug eluting stents were available for use at WFUBMC

SUMMARY:
The effectiveness, safety, and deliverability of second generation drug eluting stents (DES), including Xience V, will need to be examined in real world patients to provide the same level of evidence base and comfort that has accompanied the use of the first generation devices. Randomized clinical trials provide the fairest evaluation of outcomes by controlling for confounding patient and procedural characteristics; however, randomized clinical trials also exclude the very high risk patients that account for upwards of 80% of real world patient populations such as those at Wake Forest University Baptist Medical Center (WFUBMC).

Clinical follow-up data including non-fatal MI, all cause mortality and stent thrombosis, as well as medications compliance, of patients undergoing stent therapy including Xience V in a real world patient population will be collected at WFUBMC. Existing data for several control groups will be used to compare outcomes with Xience V including a consecutively treated bare metal stent (BMS) cohort of 1,200 patients, and a DES cohort of 1,200 patients (900 sirolimus-eluting and 300 paclitaxel-eluting) treated between April 2004 and April 2005. Patients undergoing stent therapy in the year prior to use of Xience V, and contemporaneous patients receiving non-Xience V stent therapy during Xience V use will serve as additional controls. All patient data will be de-identified using unique blinded identification codes after data collection is completed.

The null hypothesis of this study states that safety outcomes (stent thrombosis, non-fatal MI, death) with Xience V will be equivalent to historical and contemporaneous controls; effectiveness outcomes (target lesion and target vessel revascularization) with Xience V will be superior to historical and contemporaneous BMS controls, and equivalent to historical and contemporaneous DES controls; and the need for crossover to another stent type will be equal to that observed with historical DES controls. Outcomes will be reported using contemporary measures of clinical outcomes and analyzed using Cox proportional hazards survival analysis methodology. These data should provide important information on the clinical effectiveness and safety of Xience V in routine practice.

ELIGIBILITY:
Inclusion Criteria:

* percutaneous coronary intervention with stenting

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with coronary artery disease seen at WFUBMC cardiac catheterization laboratory who received percutaneous coronary intervention with placement of one or more stents
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2009-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Composite of non-fatal myocardial infarction, death, or stent thrombosis | Annual landmark

SECONDARY OUTCOMES:
Target lesion/vessel revascularization | Annual landmark

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Applegate, MD, Principal Investigator — Wake Forest University
Locations (1):
- Wake Forest University School of Medicine, Winston-Salem, North Carolina, United States